CLINICAL TRIAL: NCT02702570
Title: Committed Actions for Successful Aging
Acronym: CASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yonas E Geda, MD, Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-008490
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Brain Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CASA intervention (Other): Each participant serves as his/her own control. Measures administered before and after an intervention.
  Interventions: Behavioral: CASA

INTERVENTIONS:
Behavioral: CASA — Each participant serves as his/her own control. Measures administered before and after the behavioral intervention.

SUMMARY:
The investigators are planning to recruit approximately 30 study participants aged 50 years and older that will undergo a 4 week attention and emotion regulation intervention. The intervention systematically targets thoughts, emotions and behavior in order to promote quality of life and advance successful brain aging. The investigators will assess the feasibility of recruiting and retaining participants for an attention and emotion regulation intervention. In addition, the investigators will determine the efficacy of the intervention to enhance and promote quality of life, sustained attention, emotions, motivation and cognitive health.

DETAILED DESCRIPTION:
The CASA model is developed here in the investigators program (Geda et al) based on neuroscience and Acceptance and Commitment Therapy (ACT). The rationale for the study is that the cortico-cortical network linking the prefrontal cortex with the mesial temporal lobe is susceptible to the wear and tear of day to day life such as stress and emotional distress. The investigators hypothesize that the CASA intervention will promote emotional and cognitive health by targeting this network.

ELIGIBILITY:
Participants will be recruited from the community via advertisement in retirement communities, church, and other social gatherings. Eligible participants are cognitively normal males and females aged 50 years and older.

Inclusion criteria:

* Subject will sign approved consent form
* Male or female adults (age > 50 years of age)
* Subject will complete all of the testing and procedures

Exclusion criteria:

* Refusal to sign the approved consent form
* Refusal to complete all testing and procedures of the study
* Males and females < age of 50 years

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF quality of life questionnaire | Baseline, one year
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials. Scoring is 1-5 with 1 being either - Not at all, Very poor, Very dissatisfied, or Never. 2 being either - Not much, Poor, Dissatisfied, A little, or Seldom. 3 being either - Moderately, Neither poor nor good, Neither satisfied nor dissatisfied, A moderated amount, or Quite often. 4 being either - A great deal, Good, Satisfied, Very much, Mostly, Good, or Very often. 5 being either - Completely, Very good, Very satisfied, An extreme amount, Extremely, or Always.

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline, one year
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. The scale also includes a number of direct queries about current levels of experienced stress. The PSS was designed for use in community samples with at least a junior high school education. The questions are of a general nature and hence are relatively free of content specific to any subpopulation group. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yonas E Geda, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials